CLINICAL TRIAL: NCT04511299
Title: Impact of Fish Oil-enriched Intravenous Lipid Emulsion in Parenteral Nutrition of Phospholipid Fatty Acid Composition and Inflammatory Response in Infants After Gastrointestinal Surgery.
Brief Title: Impact of Fish Oil-enriched Lipid Emulsion on Fatty Acid and Inflammatory Response in Infants After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Principal Investigator, Meta Herdiana Hanindita, dr., Sp.A (K), MD, Pediatrician (Consultant), Dr. Soetomo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1983/105/II/2020
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Surgery
Keywords: Parenteral nutrition; Interleukin-1b; Interleukin-8; Lipid emulsion
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish oil-enriched intravenous lipid emulsion (Experimental): SMOFlipid 20%, given for 3 consecutive days with 1-4 g/kg/day.
  Interventions: Other: SMOFlipid 20%
- Standard intavenous lipid emulsion (Active Comparator): Lipofundin 20%, given for 3 consecutive days with 1-4 g/kg/day.
  Interventions: Other: Lipofundin 20%

INTERVENTIONS:
Other: SMOFlipid 20% — Fish oil-enriched intravenous lipid emulsion
  Arms: Fish oil-enriched intravenous lipid emulsion
Other: Lipofundin 20% — MCT/LCT standard intravenous lipid emulsion
  Arms: Standard intavenous lipid emulsion

SUMMARY:
This study aim to compare the impact of fish oil-enriched intravenous lipid emulsion to standard Intravenous lipid emulsion on fatty acid composition and inflammatory response (IL-1β and IL-8 levels) in infants after gastrointestinal surgery. Our hypothesis is the fish oil-enriched intravenous lipid emulsion can improve the fatty acid composition and lower the inflammatory response.

DETAILED DESCRIPTION:
This study is conducted in infants post gastrointestinal surgery that requires parenteral nutrition for at least 3 days. Subjects are classified into two groups. Group 1 received standard IVFE and group 2 received ω-3-enriched IVFE. The type of intravenous standard and omega-3-enriched fat emulsion used in this study are Lipofundin 20% and SMOFlipid 20%, respectively, both administered for three consecutive days after surgery (72 hours) in 1-4 gram/kilogram/day dosing. The inflammatory response (IL-1β and IL-8 levels) and fatty acid composition are checked from blood plasma. Blood examination is done before the surgery and 3 days after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in this study (through informed consent)
* undergo gastrointestinal surgery
* get parenteral nutrition for at least 3 days

Exclusion Criteria:

* chronic diseases
* allergic to fish, egg, soy and/or nut proteins

Ages: 1 Hour to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Fatty Acids Composition | 3 days (before surgery and after surgery)
  The percentage of fatty acid consentration from total fatty acids
Inflammatory response | 3 days (before surgery and after surgery)
  Interleukin 1b and Interleukin 8 levels

SECONDARY OUTCOMES:
Hemoglobin | 3 days (before surgery and after surgery)
  Hemoglobin value in all subjects
Leukocyte | 3 days (before surgery and after surgery)
  Leukocyte value in all subjects
C reactive Protein | 3 days (before surgery and after surgery)
  C Reactive Protein valuel in all subjects
Albumin | 3 days (before surgery and after surgery)
  Albumin value in all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Meta H Hanindita, Principal Investigator — Dr. Soetomo General Hospital
Locations (1):
- Dr. Soetomo General Hospital, Surabaya, Indonesia

IPD SHARING:
Plan to Share IPD: No